CLINICAL TRIAL: NCT03001700
Title: PRospective Study for the TrEatment of Atherosclerotic Lesions in the Superficial Femoral and/or Popliteal Arteries Using the Serranator DevicE: PRELUDE Study
Brief Title: PRospective Study for the TrEatment of Atherosclerotic Lesions in the Superficial Femoral and/or Popliteal Arteries Using the Serranator DevicE
Acronym: PRELUDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cagent Vascular LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-0109
Record Dates: First submitted 2016-12-16; First posted 2016-12-23 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Subjects will be treated with the Serranator™ Alto PTA Serration Balloon Catheter device
  Interventions: Device: Serranator™ Alto PTA Serration Balloon Catheter

INTERVENTIONS:
Device: Serranator™ Alto PTA Serration Balloon Catheter — The Serranator™ is an over-the-wire (OTW) balloon dilatation catheter designed to perform percutaneous transluminal angioplasty (PTA) for peripheral indications.

SUMMARY:
To assess preliminary safety and efficacy of the Serranator™ Alto PTA Serration Balloon Catheter in subjects with atherosclerotic peripheral artery disease of the superficial femoral and popliteal arteries.

DETAILED DESCRIPTION:
Single Arm, prospective, OUS multi-center feasibility study enrolling up to 30 subjects with superficial femoral or popliteal lesions. The study will capture acute angiographic data to compare the pre- Serranator™ inflation vs post inflation effects.

The study population will consist of subjects with claudication or ischemic rest pain, with de novo or non-stented restenotic lesions in femoropopliteal arteries having lesion length less than or equal to 10 cm, total occlusion up to 6 cms in length and reference vessel diameter of 4 mm to 6 mm, inclusive.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of >18 years old.
2. Women of child bearing potential must have a negative pregnancy test within 7 days of index procedure.
3. Subject or subject's legal representative has been informed of the nature of the study, agrees to participate and comply with all follow-up visits and has signed the consent form.
4. Resting ABI -< 0.9.
5. Subject is eligible for standard surgical repair in target limb if necessary.
6. Subject has Rutherford Clinical Category 2,3, or 4
7. Estimated life expectancy > 1 year.

Angiographic Inclusion Criteria:

1. Lesion(s) located within the SFA and or popliteal arteries.
2. Target lesion(s) has stenosis >70% by visual assessment.
3. Reference vessel diameter is between 4.0mm and 6.0mm, inclusive.
4. One long or multiple serial lesions that are up to 10 cms, (total occlusions up to 6cm) in length that can be covered by a single balloon.
5. De-novo, or non-stented re-stenotic lesions
6. At least one below the knee artery patent to the ankle.
7. Successful treatment of iliac inflow stenosis to the target limb. Stenosis can be treated during the same procedure using standard angioplasty and or stenting but use of atherectomy is excluded. The inflow lesion(s) must be treated first, prior to consideration of treatment of the target lesion. Subject can be enrolled if the inflow lesion(s) are treated and results in <30% residual stenosis and no evidence of embolization or significant complications.

Exclusion Criteria:

1. Rutherford Clinical Category 1, 5 or 6.
2. Previously implanted ipsilateral femoral or popliteal stent.
3. Evidence of aneurysm or acute thrombus in the target vessel.
4. Subjects with previous bypass surgery in lower target extremity.
5. Planned major amputation (above the ankle) of either limb.
6. Subject has significant stenosis or occlusion of inflow tract not successfully treated (>30% residual stenosis and/or significant complication of the procedure).
7. History of any open surgical procedure within the past 30 days.
8. Planned endovascular or vascular surgery procedure within 14 days prior to the ATK procedure, except to treat the inflow vessels on the day of the procedure, or within the next 30 days after the ATK procedure on the target limb.
9. Subject has an allergy to contrast medium that cannot be pretreated.
10. Episode of acute limb ischemia within past 30 days.
11. Subject has systemic infection with positive blood cultures/ bacteremia within one week.
12. Subject has a hypercoagulable disorder
13. Subject in whom antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated.
14. Myocardial infarction within 30 days prior to enrollment.
15. History of stroke or TIA within 90 days prior to enrollment.
16. Subject has acute or chronic renal disease (e.g., as measured by a serum creatinine of >2.5 mg/dL or >220 umol/L).
17. Subject is pregnant or breastfeeding.
18. Subject is participating in another research study of a device, medication, which could, in the opinion of the investigator, affect the results of this study.
19. Subject has other medical, social or psychological problems that in the opinion of the investigator would preclude them from receiving this treatment and the procedures and or participating in evaluations pre- and post-treatment.
20. Thrombolysis of the target vessel within 72 hours prior to the index procedure, where complete resolution of the thrombus was not achieved.
21. Known allergies to both antiplatelet agents, aspirin, or heparin.
22. History of neutropenia, coagulopathy, or thrombocytopenia that was unexplained or is considered to be at risk for reoccurrence.
23. Platelet count less than 80,000/μL,
24. Subject requires general anesthesia for the procedure.
25. Subject requires dialysis.

Angiographic Exclusion Criteria:

1. Chronic Total Occlusions (CTO) > 6cm in length
2. Acute Total Occlusions; evidence of acute thrombus formation by angiography
3. Severe calcification of target lesion described as circumferential calcium and >50% of lesion length.
4. Sub-intimal access required
5. Inability to cross the lesion with a guidewire
6. Atherectomy in the target lesion, target artery or for inflow treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the technical feasibility of using the Serranator™ Alto PTA Serration Balloon Catheter during the endovascular treatment of critical SFA or popliteal artery lesions. | Through Study Completion, approximately 6 months

SECONDARY OUTCOMES:
OCT and/or IVUS imaging post use of the Serranator to document evidence of vessel wall serrations in a sub-set of up to 10 subjects. | Through Study Completion, approximately 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- Medizinische Universtität Graz, Graz, Austria
- Auckland City Hospital, Auckland, Grafton, New Zealand
- Poland (2):
  - Polsko-Amerykańskie Kliniki Serca PAKS Małopolskie Centrum Sercowo Naczyniowe, Chrzanów
  - Szpital Uniwersytecki w Krakowie Pracownia Angiografii Oddział Angiologii, Krakow

IPD SHARING:
Plan to Share IPD: No